CLINICAL TRIAL: NCT05252611
Title: The Validity and Reliability of the Turkish Version of the Chronic Pain Acceptance Questionnaire-8
Brief Title: The Validity and Reliability of the Turkish Version of the CPAQ-8
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Kivanc Menekseoglu, Principal Investigator, Istanbul University
Other Study IDs: 2019/58
Record Dates: First submitted 2022-02-12; First posted 2022-02-23 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Fibromyalgia; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Turkish version of the Chronic Pain Acceptance Questionnaire-8 (CPAQ-8) — The aim of this study is to test the validity of the Turkish version of the Chronic Pain Acceptance Questionnaire-8 (CPAQ-8).

SUMMARY:
Acceptance of chronic pain is becoming an increasingly important issue in the field of pain management. Many researchers argue that patients who accept pain better function better both physically and psychologically. In many countries, the Chronic Pain Acceptance Questionnaire - 8 (CPAQ-8) has been frequently validated and used to measure the pain acceptance of patients with chronic pain.1 However, the CPAQ-8 has not yet been introduced and validated in Turkey. In this study, we aimed to translate the English version of CPAQ-8 into Turkish, make correct cross-cultural adaptations, and validate the psychometric properties of the Turkish version of CPAQ-8 by testing it in Turkish fibromyalgia patients.

DETAILED DESCRIPTION:
Chronic pain is an undesirable condition that affects a large part of the society and increases the psychological and economic burden of the population it affects. Psychological variables are known to be strong in the perception of pain and especially cause patients to avoid activity in order to reduce pain. Individuals prefer to avoid painful experiences when they are worn out in repetitive attempts to control and prevent pain, which ultimately causes pain to become more dominant and destructive, and activities that are valuable to the individual are neglected.1 At this point, accepting pain can be seen as the antithesis of avoiding painful experiences. Acceptance of pain is a strong predictor of low disability in chronic pain.2 The Chronic Pain Acceptance Questionnaire (CPAQ) represents one of the ways in which pain acceptance is functionalized and measured in the context of chronic pain. The short form of CPAQ, CPAQ-8, was developed and validated recently and shows the same factor structure, reliability and validity as the 20-factor version. Given that psychometric testing is an incremental process, further evaluation of the questionnaire is desirable, including test-retest reliability and replication of results reported by Fish et al.

ELIGIBILITY:
Inclusion Criteria:

* Patients who applied to our physical medicine and rehabilitation outpatient clinic,
* Agreed to participate in the study, were over the age of 18,
* Had at least primary school education, were diagnosed with fibromyalgia syndrome according to the 2016 American College of Rheumatology (ACR) criteria,
* Could speak and communicate in Turkish were included in the study.

Exclusion Criteria:

* Those who did not agree to participate in the study,
* <18 years old, and could not communicate in Turkish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to our physical medicine and rehabilitation outpatient clinic, agreed to participate in the study, were over the age of 18, had at least primary school education, were diagnosed with fibromyalgia syndrome according to the 2016 American College of Rheumatology (ACR) criteria, and could speak and communicate in Turkish were included in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 01.01.2020-31.12.2021
  The Fibromyalgia Impact Questionnaire was used to measure patients' symptom severity and functional status. There are 10 items in the FIQ; each item gets a score between 0-10. The first item questions the ability to perform activities of daily living with 11 questions. Other items question general well-being, ability to work, and symptoms of pain, fatigue, stiffness, anxiety, and depression. The score range is 0 to 100; higher scores indicate severe disease.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | 01.01.2020-31.12.2021
  Hospital Anxiety and Depression Scale (HADS) consists of 14 items. It is designed to assess the severity of anxiety and depression in patients.Each item is scored between 0-3; higher scores indicate more anxiety or depression.
Tampa Scale of Kinesiophobia | 01.01.2020-31.12.2021
  Tampa Scale of Kinesiophobia (TSK) is a 17 item self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. . Scoring ranges from 1 to 4 points for each item, with higher scores indicating greater fear of injury.
Brief Pain Inventory | 01.01.2020-31.12.2021
  Brief Pain Inventory consists of four questions about the severity of pain and seven questions about its effect on daily functions. The inventory assesses an individual's walking, exercise, sleep, emotional state, general activity status, social relations, and joy in the last 24 hours. Each item gets scored between 0 and 10, ; higher scores indicate severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet K Menekşeoğlu, Principal Investigator — Kanuni Sultan Süleyman Research and Training Hospital
Locations (1):
- Ahmet Kıvanç Menekşeoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fish RA, Hogan MJ, Morrison TG, Stewart I, McGuire BE. Willing and able: a closer look at pain Willingness and Activity Engagement on the Chronic Pain Acceptance Questionnaire (CPAQ-8). J Pain. 2013 Mar;14(3):233-45. doi: 10.1016/j.jpain.2012.11.004. PMID 23452647
- [Result] Fish RA, McGuire B, Hogan M, Morrison TG, Stewart I. Validation of the chronic pain acceptance questionnaire (CPAQ) in an Internet sample and development and preliminary validation of the CPAQ-8. Pain. 2010 Jun;149(3):435-443. doi: 10.1016/j.pain.2009.12.016. Epub 2010 Feb 25. PMID 20188472
- [Result] Kleinebrecht J, Degenhardt KH, Franz J, Schneider G. Variability of limb malformations induced by 5-fluoro-2'-deoxycytidine in mice. Teratology. 1972 Jun;5(3):295-301. doi: 10.1002/tera.1420050304. No abstract available. PMID 5032639